CLINICAL TRIAL: NCT03813147
Title: A Feasibility Trial of MLN4924 (Pevonedistat, TAK 924) Given in Combination With Azacitidine, Fludarabine, and Cytarabine, in Children, Adolescents, and Young Adults With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Pevonedistat, Azacitidine, Fludarabine Phosphate, and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00215; NCI-2019-00215 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1712 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1712 (Other: CTEP)
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Cytarabine; fludarabine phosphate; Methotrexate; merphos; pevonedistat; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cytarabine, azacitidine, pevonedistat, fludarabine) (Experimental): Patients receive cytarabine intrathecally on day 0 at least 24 hours prior to the start of each cycle. Patients then receive azacitidine IV over 15 minutes QD on days 1-5, pevonedistat IV over 60 minutes on days 1, 3, and 5, and fludarabine phosphate IV over 30 minutes QD and cytarabine IV over 1-3 hours QD on days 6-10. Patients with CNS2 or CNS3 receive cytarabine intrathecally or methotrexate intrathecally, hydrocortisone intrathecally, and cytarabine intrathecally on days 8 and 11-34. Cycles continue for 35 days in the absence of disease progression or unacceptable toxicity. Patients with stable or greater with non-hematologic toxicities probably or definitely related to pevonedistat may receive an additional cycle of treatment.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Fludarabine Phosphate; Drug: Methotrexate; Drug: Pevonedistat; Drug: Therapeutic Hydrocortisone

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Cytarabine — Given intrathecally and IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Methotrexate — Given intrathecally
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924
Drug: Therapeutic Hydrocortisone — Given intrathecally
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid

SUMMARY:
This phase I trial studies the side effects and how well pevonedistat, azacitidine, fludarabine phosphate, and cytarabine work in treating patients with acute myeloid leukemia or myelodysplastic syndrome that has come back (relapsed) or has not responded to treatment (refractory). Pevonedistat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as azacitidine, fludarabine phosphate, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) and pevonedistat may work better in treating patients with acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the tolerability and feasibility of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine phosphate (fludarabine), and cytarabine re-induction for pediatric patients with recurrent/refractory acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS).

II. To define and describe the toxicities of MLN4924 (pevonedistat) when given in combination with azacitidine, fludarabine, and cytarabine to pediatric patients with relapsed/refractory AML and MDS.

III. To characterize the pharmacokinetics of MLN4924 (pevonedistat) in children with recurrent or refractory AML and MDS.

SECONDARY OBJECTIVE:

I. To describe the antitumor activity of MLN4924 (pevonedistat) in combination with azacitidine, fludarabine, and cytarabine within the confines of a feasibility study.

EXPLORATORY OBJECTIVES:

I. To describe the effect of MLN4924 (pevonedistat) administered on this schedule on messenger ribonucleic acid (mRNA) transcript levels of genes known to be induced by MLN4924 (pevonedistat) mediated NEDD8 activating enzyme (NAE) inhibition.

II. To describe the effect of MLN4924 (pevonedistat) on NEDDylation of proteins in the NEDD8 pathway that are likely to be affected by NAE inhibition with MLN4924 (pevonedistat).

OUTLINE:

Patients receive cytarabine intrathecally on day 0 at least 24 hours prior to the start of each cycle. Patients then receive azacitidine intravenously (IV) over 15 minutes once daily (QD) on days 1-5, pevonedistat IV over 60 minutes on days 1, 3, and 5, and fludarabine phosphate IV over 30 minutes QD and cytarabine IV over 1-3 hours QD on days 6-10. Patients with central nervous system (CNS)2 or CNS3 receive cytarabine intrathecally or methotrexate intrathecally, hydrocortisone intrathecally, and cytarabine intrathecally on days 8 and 11-34. Cycles continue for 35 days in the absence of disease progression or unacceptable toxicity. Patients with stable or greater with non-hematologic toxicities probably or definitely related to pevonedistat may receive an additional cycle of treatment.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of AML at the original diagnosis. Patients must have one of the following:

  * Recurrent disease in >= 1st relapse with >= 5% blasts in the bone marrow (M2/M3) marrow OR immunophenotypic evidence of disease with >= 0.1% blasts detected by flow cytometry, OR evidence of recurrent cytogenetic or molecular abnormalities consistent with relapse, with or without extramedullary disease
  * Refractory AML is defined as >= 5% blasts in the bone marrow (M2/M3) after >= 2 induction attempts (i.e., 2 cycles of chemotherapy)
  * Patients with advanced MDS, including MDS that has progressed to AML, and have experienced relapse or are refractory after >= 1 course of induction therapy, are eligible
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea, for patients not receiving standard maintenance therapy. Additionally, patients must have recovered from all acute toxic effects of prior therapy

      * NOTE: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without traumatic brain injury [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor leukocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular Therapy: >= 30 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 42 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial brain metastases (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131 iodine [I]-metaiodobenzylguanidine [MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to MLN4924 (pevonedistat)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months; 0.4 (male and female)
  * 6 months to < 1 year; 0.5 (male and female)
  * 1 to < 2 years; 0.6 (male and female)
  * 2 to < 6 years; 0.8 (male and female)
  * 6 to < 10 years; 1 (male and female)
  * 10 to < 13 years; 1.2 (male and female)
  * 13 to < 16 years; 1.5 (male) and 1.4 (female)
  * >= 16 years; 1.7 (male) and 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< upper limit of normal (ULN) for age
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN. For the purpose of this study, the ULN for serum glutamate pyruvate transaminase (SGPT) is 45 U/L
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by echocardiogram or radionuclide angiogram
* No ventricular or supraventricular arrhythmia on electrocardiogram (EKG)
* Prolonged rate corrected QT (QTc) interval < 500 msec
* Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest)
* International normalized ratio (INR) =< 1.5
* Hemoglobin > 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use 1 highly effective and 1 additional effective (barrier) method of contraception at the same time for the duration of study therapy and for 4 months after the completion of MLN4924 (pevonedistat) administration. True abstinence, when this is in line with the preferred and usual lifestyle of the subject, is acceptable. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception
* Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible (except hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy)
* Anti-GVHD agents post-transplant: Patients who are receiving cyclosporine, tacrolimus or other systemic agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial. Topical immunosuppressive agents (e.g. topical steroids) are allowed. Physiologic replacement of hydrocortisone is allowed
* Patients who are taking drugs that are strong CYP3A4 inducers and cannot be switched to alternative drugs 14 days prior to enrollment are not eligible. Strong inducers of CYP34 are not permitted during the study
* Patients with known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection are not eligible. NOTE: Patients who have isolated positive hepatitis B core antibody (i.e. in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* Patients with known hepatic cirrhosis or severe pre-existing hepatic impairment are not eligible
* Patients with uncontrolled high blood pressure (i.e., >= 99% for age) are not eligible
* Patients with any of the following diagnoses:

  * Acute promyelocytic leukemia
  * Down syndrome
  * Juvenile myelomonocytic leukemia
* Patients who have a documented active uncontrolled infection are not eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as the study agent
* Patients with human immunodeficiency virus (HIV) are not eligible unless they meet all of the following criteria:

  * CD4 count > 350 cell/mm^3
  * Undetectable viral load
  * Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s) are not eligible
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s) are not eligible

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine G Tarlock, Principal Investigator — COG Phase I Consortium
Locations (19):
- United States (19):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were treated at the 20 mg/m2 dosing. An initial 6 patients were treated in this stratum to ensure this dose was feasible with the backbone therapy and then an additional 6 patients were treated in the PK stratum at this same dose to gain additional PK data.
Groups:
- Stratum 1 With 20 mg/m^2; PK With 20 mg/m^2: Treatment (cytarabine, azacitidine, pevonedistat, fludarabine)
Period: Overall Study
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Started | 6 | 6
Completed | 0 | 1
Not Completed | 6 | 5
Not completed — Lack of Efficacy | 4 | 4
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 9.5 [3 to 17] | 16.5 [1 to 21] | 13 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities of MLN4924 (Pevonedistat)
Description: Frequency of patients with dose limiting toxicity in the first cycle of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level among patients in the dose escalation cohort.
Time Frame: Up to 35 days
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

2. Primary Outcome: Number of Participants With Adverse Events Attributable to MLN4924 (Pevonedistat)
Description: Frequency of patients with at least one grade 3 adverse event at least possibly attributable to MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level.
Time Frame: Up to 70 days
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (Range) of the area under the plasma concentration versus time curve of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level measured pre-dose, end of infusion, 4-6 hours, and 24 hours post-dose infusion on Days 1 and 5.
Time Frame: Up to 5 days
Population: All eligible patients
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 1004.9 [637.8 to 1381.4] | 1047.4 [727.6 to 1362.6]

4. Primary Outcome: Total Plasma Clearance of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (Range) of the total plasma clearance of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level measured pre-dose, end of infusion, 4-6 hours, and 24 hours post-dose infusion on Days 1 and 5.
Time Frame: Up to 5 days
Population: All eligible patients
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
L/h/m^2 | 20.1 [14.4 to 31.4] | 19.2 [14.8 to 27.5]

5. Primary Outcome: Elimination Half-life of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (Range) of the elimination half-life of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level measured pre-dose, end of infusion, 4-6 hours, and 24 hours post-dose infusion on Days 1 and 5.
Time Frame: Up to 5 days
Population: All eligible patients
Measure: Median (Full Range); unit: Hour
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
Hour | 4.7 [1.9 to 5.2] | 5.5 [3.8 to 6.1]

6. Primary Outcome: Maximum Concentration of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (Range) of the maximum concentration of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level measured pre-dose, end of infusion, 4-6 hours, and 24 hours post-dose infusion on Days 1 and 5.
Time Frame: Up to 5 days
Population: All eligible patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
ng/mL | 248.5 [168.0 to 362.0] | 213 [132.0 to 400.0]

7. Primary Outcome: Maximum Time to Concentration of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (Range) of the maximum time to concentration of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level measured pre-dose, end of infusion, 4-6 hours, and 24 hours post-dose infusion on Days 1 and 5.
Time Frame: Up to 5 days
Population: All eligible patients
Measure: Median (Full Range); unit: Hour
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
Hour | 1.2 [1.0 to 1.2] | 1.1 [1.0 to 1.5]

8. Secondary Outcome: Number of Participants With Antitumor Activity of MLN4924 (Pevonedistat)
Description: Frequency of participants with best overall response by dose level of PR or CR for MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction Per Response Evaluation Criteria for CR (M1 bone marrow (< 5% blasts) with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral blood counts (ANC > 1000/uL and platelet count > 100,000/uL), CRp (M1 bone marrow (< 5% blasts) and no evidence of circulating blasts or extramedullary disease and with recovery of ANC > 1000/uL and platelet transfusion independence), CRi (M1 bone marrow (<5% blasts) and no evidence of circulating blasts or extramedullary disease and with ANC < 1000/uL or platelet count < 100,000/uL without platelet transfusion independence), or PR (M2 marrow status (> 5% or < 25% blasts cells) and at least 50% decrease in bone marrow blast percent from baseline.
Time Frame: Up to 1 year
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

9. Other Pre Specified Outcome: Messenger Ribonucleic Acid (mRNA) Transcript Levels of MLN4924 (Pevonedistat) Added to the 3-drug Backbone of Azacitidine (Aza), Fludarabine, and Cytarabine Re-induction for Pediatric Patients With Recurrent/Refractory AML and MDS
Description: Median (IQR) transcript levels of MLN4924 (pevonedistat) added to the 3-drug backbone of azacitidine (aza), fludarabine, and cytarabine re-induction for pediatric patients with recurrent/refractory AML and MDS by dose level.
Time Frame: Up to 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Stratum 1 With 20 mg/m^2 | PK With 20 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 20 mg/m^2 (N=6) | PK With 20 mg/m^2 (N=6)
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Allergic reaction (Immune system disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Fever (General disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
GGT increased (Investigations) | 1 | 0
Heart failure (Cardiac disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Irritability (Psychiatric disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 6
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 6 | 6
Obesity (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 6 | 6
Proteinuria (Renal and urinary disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 6 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 20 mg/m^2 (N=6) | PK With 20 mg/m^2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Agitation (Psychiatric disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 5 | 4
Alkaline phosphatase increased (Investigations) | 1 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 6
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 3
Blurred vision (Eye disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Cardiac disorders - Other, (Cardiac disorders) | 1 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cholesterol high (Investigations) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Creatinine increased (Investigations) | 1 | 1
Depression (Psychiatric disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Edema face (General disorders) | 1 | 1
Edema limbs (General disorders) | 2 | 2
Edema trunk (General disorders) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye disorders - Other, (Eye disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 4 | 4
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 3 | 3
Floaters (Eye disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
GGT increased (Investigations) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorders - Other, (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hematoma (Vascular disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Hemoglobin increased (Investigations) | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Hepatobiliary disorders - Other, (Hepatobiliary disorders) | 1 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Hypotension (Vascular disorders) | 4 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
INR increased (Investigations) | 1 | 1
Immune system disorders - Other, (Immune system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Investigations - Other, (Investigations) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 2
Malaise (General disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1
Movements involuntary (Nervous system disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4
Neck edema (General disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Phlebitis infective (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Psychiatric disorders - Other, (Psychiatric disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary valve disease (Cardiac disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Renal and urinary disorders - Other, (Renal and urinary disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Scleral disorder (Eye disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 2
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 2 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1
Tooth discoloration (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 3
Weight loss (Investigations) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03813147/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03813147/ICF_001.pdf